CLINICAL TRIAL: NCT00339898
Title: Prospective Evaluation of the Prognostic Relevance of PCR Positivity in Blood and Bone Marrow in Non-Metastatic Ewings Sarcoma
Brief Title: Prognostic Value of a Positive RT-PCR Test in Patients With Ewing Sarcoma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904135; 04-C-N135; NCT00899236 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-01-13

CONDITIONS: Non-Metastatic Ewings Sarcoma
Keywords: Minimal Residual Disease; Ewings Sarcoma
MeSH Terms: conditions — Neoplasm, Residual; Sarcoma, Ewing

SUMMARY:
This study will determine whether the results of a test called reverse transcriptase-polymerase chain reaction (RT-PCR) correlate with clinical outcomes in patients with Ewing sarcoma, and if they can be used to help identify patients at high risk for metastasis (spread of the cancer beyond the original site).

This is a companion study to another NCI trial (AEWS0031), which is examining the effectiveness of an intensified chemotherapy regimen for patients with Ewing sarcoma. The primary purposes of AEWS0031 are to determine: 1) if chemotherapy given every 2 weeks can cure more patients with Ewing sarcoma and similar tumors than chemotherapy given every 3 weeks; and 2) if certain biological characteristics of these tumors can predict how well the chemotherapy will work.

Many, but not all, patients with Ewing sarcoma that has not metastasized can be cured with standard radiation, surgery, and chemotherapy treatment. Most patients whose tumors have spread, however, are not cured with standard treatment. A goal of future therapy is to identify patients at highest risk for metastasis so that they can be given more intensive therapy, and, conversely, patients at lower risk of relapse can receive less toxic treatment.

Patients enrolled in AEWS0031 are eligible for this companion study. No additional procedures re required; RT-PCR testing will be performed on blood and bone marrow samples collected for AEWS0031.

...

DETAILED DESCRIPTION:
BACKGROUND: Clinical evidence for metastatic disease at the time of diagnosis is an indicator of poor prognosis in Ewing's sarcoma. Patients with non-metastatic disease at presentation are thought to have a better prognosis than those with metastatic disease. Unfortunately, patients who appear non-metastatic at presentation may relapse after initiating or completing standard therapy for Ewing's sarcoma. Evidence of metastatic disease may be determined by radiographic studies and biopsy of potential site(s) of disease. It is possible to identify submicroscopic Ewing's sarcoma cells in blood and bone marrow, yet the prognostic value of this finding is unclear.

OBJECTIVES: To determine the incidence of RT PCR positivity in the blood and bone marrow of patients enrolled on COG AEWS0031 and to correlate the clinical outcome with RT PCR positivity.

ELIGIBILITY: Concurrent enrollment on COG AEWS0031.

DESIGN: This is a Companion Biology Study, enrolling approximately 500 patients. All specimens will be evaluated for translocations, it is anticipated that approximately 30% of specimens will have RT PCR positivity. Specimens are collected at the time of diagnosis, prior to cycle 2 chemotherapy, prior to initiation of local control, and at the end of therapy/follow up. Batched specimens are provided to the NIH by the Cooperative Human Tissue Network (CHTN). Following the completion of the COG trial and appropriate follow up periods, RT PCR positivity will be compared with clinical outcome to determine prognostic value.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients enrolled on COG AEWS0031 are eligible for this study.

EXCLUSION CRITERIA:

Patients who were enrolled but from whom samples were not obtained will not be enrolled on this study.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 414 (Actual)
Dates: Start 2004-03-12; Study Completion 2015-01-13

CONTACTS AND LOCATIONS:
Overall Officials: Crystal L Mackall, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Grier HE, Krailo MD, Tarbell NJ, Link MP, Fryer CJ, Pritchard DJ, Gebhardt MC, Dickman PS, Perlman EJ, Meyers PA, Donaldson SS, Moore S, Rausen AR, Vietti TJ, Miser JS. Addition of ifosfamide and etoposide to standard chemotherapy for Ewing's sarcoma and primitive neuroectodermal tumor of bone. N Engl J Med. 2003 Feb 20;348(8):694-701. doi: 10.1056/NEJMoa020890. PMID 12594313
- [Background] West DC, Grier HE, Swallow MM, Demetri GD, Granowetter L, Sklar J. Detection of circulating tumor cells in patients with Ewing's sarcoma and peripheral primitive neuroectodermal tumor. J Clin Oncol. 1997 Feb;15(2):583-8. doi: 10.1200/JCO.1997.15.2.583. PMID 9053480
- [Background] Pfleiderer C, Zoubek A, Gruber B, Kronberger M, Ambros PF, Lion T, Fink FM, Gadner H, Kovar H. Detection of tumour cells in peripheral blood and bone marrow from Ewing tumour patients by RT-PCR. Int J Cancer. 1995 Apr 21;64(2):135-9. doi: 10.1002/ijc.2910640211. PMID 7542227